CLINICAL TRIAL: NCT02861391
Title: Evaluation of the Safety and Efficacy of CO2 Acupulse Laser Treatment on Women With Urinary Stress Incontinence.
Brief Title: Evaluation of the Safety and Efficacy of Carbon Dioxide (CO2) Acupulse Laser Treatment on Urinary Stress Incontinence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Dr. Roy Lauterbach, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0205-16-RMB
Record Dates: First submitted 2016-07-25; First posted 2016-08-10 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Exposure Laser

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 AcuPulse Laser treatment (Experimental): Subjects with USI as diagnosed by cough test intended to receive 3 laser treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.
  Interventions: Device: CO2 AcuPulse Laser
- Sham laser treatment (Sham Comparator): Subjects with USI as diagnosed by cough test intended to receive 3 sham treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.
  Interventions: Device: Sham Laser

INTERVENTIONS:
Device: CO2 AcuPulse Laser — Each subject will receive 3 laser treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.
  Arms: CO2 AcuPulse Laser treatment
Device: Sham Laser — Each subject will receive 3 sham treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.
  Arms: Sham laser treatment

SUMMARY:
The study is intended to assess the safety and efficacy of CO2 AcuPulse laser treatment in patients with stress urinary incontinence (SUI). Eligible subjects will either receive 3 laser or sham treatment sessions, 4 weeks apart and 4 Follow Up visits, at 1, 3, 6, and 12 months following the last treatment.

DETAILED DESCRIPTION:
Following a screening visit, eligible subjects will be enrolled into the study. Eligibility will be decided depending on the level of SUI the patient has. Each subject will receive either 3 laser or sham treatments 4 weeks apart and 4 Follow Up visits, at 1, 3, 6, and 12 months following the last treatment.

Further demographic information and patient history will be obtained from the subjects' electronical files.

ELIGIBILITY:
Inclusion Criteria:

* Negative urine culture.
* Positive cough test.
* Normal Papanicolaou (PAP) test from the past 3 years.

Exclusion Criteria:

* signs, symptoms or validated test results indicating possible urgency urinary incontinence or mixed urinary incontinence.
* Overactive bladder.
* Previous bulking injections.
* Previous transvaginal mesh implant.
* Previous surgery for stress urinary incontinence.
* Presence of pelvic organ prolapse.
* Presence of an active or recurring genital infection or urinary tract infection.
* Previous laser-based or other energy-based treatments for gynecological indications.
* Vaginal bleeding of unknown reason.
* Pregnancy.
* Current pelvic floor physiotherapy.
* Current treatment with local or systemic hormone replacement therapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Pad weight test. | 15 months from recruitment.
  Pad weight results in grams.

SECONDARY OUTCOMES:
Urinary distress index 6 questionnaire. | 15 months from recruitment.
  Total questionnaire score.
Pelvic Organ Prolapse/Urinary Incontinence Sexual questionnaire. | 15 months from recruitment.
  Total questionnaire score.
International Consultation of Incontinence questionnaire. | 15 months from recruitment.
  Total questionnaire score.
Cough test | 15 months from recruitment.
  cough test results.
Visual analogue scale. | 15 months from recruitment.
  Pain rated with the visual analogue score.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No